CLINICAL TRIAL: NCT06919965
Title: A Phase 3, Randomized, Open-label, Multicenter Study Evaluating the Efficacy and Safety of TAR-210 Erdafitinib Intravesical Delivery System Versus Investigator's Choice of Intravesical Chemotherapy in Participants With High-risk Non-muscle-invasive Bladder Cancer With Susceptible FGFR Alterations Who Had Received Intravesical Bacillus Calmette-Guérin (BCG)
Brief Title: A Study to Evaluate TAR-210 Versus Intravesical Chemotherapy Treatment in Participants With High Risk Non-Muscle-Invasive Bladder Cancer
Acronym: MoonRISe-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 42756493BLC3005; 42756493BLC3005 (Other: Janssen Research & Development, LLC); 2024-519493-39-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Non-Muscle Invasive Bladder Neoplasms
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — erdafitinib; Mitomycin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: TAR-210 (Experimental): Participants in Group A will have TAR-210 inserted in the bladder on Day 1. TAR-210 will be inserted over a treatment duration of approximately 2 years.
  Interventions: Drug: TAR-210
- Group B: Mitomycin C (MMC) or Gemcitabine (Active Comparator): Participants in Group B will receive intravesical mitomycin C (MMC) or gemcitabine (investigator's choice) once weekly for 4 to 6 induction doses followed by maintenance dosing once monthly for up to 1 year. An optional second year of additional maintenance can be added at the investigator's discretion.
  Interventions: Drug: Mitomycin C; Drug: Gemcitabine

INTERVENTIONS:
Drug: TAR-210 — TAR-210 will be administered intravesically.
  Other Names: JNJ-42756493
  Arms: Group A: TAR-210
Drug: Mitomycin C — MMC will be administered intravesically.
  Arms: Group B: Mitomycin C (MMC) or Gemcitabine
Drug: Gemcitabine — Gemcitabine will be administered intravesically.
  Arms: Group B: Mitomycin C (MMC) or Gemcitabine

SUMMARY:
The main purpose of this study is to compare the disease-free survival (the length of time after randomization that a participant survives without any signs or symptoms of the cancer returning, or progressing) between Bacillus Calmette-Guérin (BCG) treated participants receiving treatment with TAR-210 versus investigator's choice of intravesical chemotherapy for treatment of high-risk non-muscle-invasive bladder cancer (HR-NMIBC).

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed diagnosis by local pathology of papillary-only HR-NMIBC (defined as high-grade Ta or any T1, no CIS). Mixed histology tumors are allowed if urothelial differentiation is predominant. However, neuroendocrine, and small cell variants will be excluded
* Have a susceptible fibroblast growth factor receptor (FGFR) mutation or fusion either by urine testing or tumor tissue testing (from TURBT tissue) as determined by central or local testing
* All visible tumor completely resected prior to randomization. Urine cytology must not be positive or suspicious for high grade UC before randomization. For participants with lamina propria invasion (T1) on the screening biopsy/TURBT, muscularis propria must be present to rule out MIBC
* Participants must have had either: a. Adequate Induction (5 of 6 doses) and either 2 of 3 doses of Maintenance or 2 of 6 doses of second Induction of BCG with high-grade T1 disease at first disease assessment after induction or high-grade Ta/any T1 disease within 6 months after last BCG (BCG-unresponsive population); b. had adequate induction (5 or 6 doses) with or without maintenance BCG with high-grade Ta/any T1 disease within 12 months after last BCG excluding BCG-unresponsive (BCG-experienced population); or c. been unable to complete an induction course of BCG with at least 5 doses due to grade >= 2 toxicity requiring BCG discontinuation (BCG intolerant population)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status Grade of 0, 1, or 2
* Must be ineligible for or refusing radical cystectomy (RC)

Exclusion criteria:

* Presence of CIS at any point from time of diagnosis of papillary-only HR-NMIBC recurrence to randomization. Additionally, presence or history of histologically confirmed, muscle-invasive, locally advanced, nonresectable, or metastatic urothelial carcinoma (that is [i.e.], T2, T3, T4, N+, and/or M+)
* Active malignancies (i.e., progressing or requiring treatment change in the last 24 months) other than the disease being treated under study. Allowed recent second or prior malignancies: a. Any malignancy that was not progressing nor requiring treatment change in the last 12 months; b. Malignancies treated within the last 12 months and considered at very low risk for recurrence for example (e.g.): non-melanoma skin cancers (treated with curative therapy or localized melanoma treated with curative surgical resection alone), non-invasive cervical cancer, breast cancer (adequately treated lobular CIS or ductal CIS, localized breast cancer and receiving antihormonal agents), localized prostate cancer ([N0, M0] with a Gleason score less than or equal to [<=] 7a, treated locally only [radical prostatectomy/radiation therapy/focal treatment]) and other malignancy that is considered at minimal risk of recurrence
* Presence of any bladder or urethral anatomic feature that, in the opinion of the investigator, may prevent the safe placement, indwelling use, or removal of TAR 210
* A history of clinically significant polyuria with recorded 24 hour urine volumes greater than (>) 4,000 milliliters (mL)
* Indwelling catheters are not permitted; however, intermittent catheterization is acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2028-04-06 (Estimated); Study Completion 2032-03-16 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) | Up to 5 years
  DFS is measured as the time from randomization to the date of the first recurrence of HR-NMIBC (high-grade Ta, any T1 or carcinoma in situ [CIS]), progression, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to 5 years
  RFS is measured as the time from randomization to the date of the first recurrence of HR-NMIBC (high-grade Ta, any T1, or CIS), or death due to any cause, whichever occurs first.
Time to Next Intervention (TTNI) | Up to 5 years
  TTNI (i.e., transurethral resection of bladder tumor [TURBT], radical cystectomy [RC], radiation therapy [RT], or chemotherapy) is measured as the time from randomization to the date of next intervention (localized or systemic) for the treatment of urothelial carcinoma (UC).
Time to Disease Worsening (TTDW) | Up to 5 years
  TTDW is measured as the time from randomization to the date of cystectomy, systemic therapy, or radiation therapy, whichever occurs first.
Time to Progression (TTP) | Up to 5 years
  TTP is measured as the time from randomization to the date of first documented evidence of disease progression (i.e., progression to muscle-invasive bladder cancer [MIBC] [T greater than or equal to {>=} 2], lymph node [N+], or distant disease [M+]), or death due to disease progression, whichever occurs first.
Overall Survival (OS) | Up to 5 years
  OS is defined as the time from randomization to death due to any cause.
Number of Participants with Adverse Events (AEs) According to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | Up to 5 years
  Number of participants with AEs by severity grade as assessed by CTCAE version 5.0 will be reported. Grade refers to the severity of AE as follows: Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe; Grade 4- Life-threatening; Grade 5- Death related to adverse event.
Number of Participants With Change from Baseline in Laboratory Abnormalities | Up to 5 years
  Number of participants with change from baseline in laboratory abnormalities (hematology, serum chemistry and urine analysis) will be reported.
Number of Participants With Change from Baseline in Vital Signs Abnormalities | Up to 5 years
  Number of participants with change from baseline in vital signs (temperature, pulse/heart rate, respiratory rate and blood pressure) will be reported.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire (EORTC QLQ)-C30 Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and 96
  EORTC QLQ-C30 is a 30-item questionnaire for evaluating the health-related quality of life (HRQoL) of participants participating in cancer clinical studies. It includes 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea or vomiting), a global health status or HRQoL scale and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Ratings for each item range from 1 (not at all) to 4 (very much). Higher scores indicate greater functioning, better global health status, or more severe symptoms.
Change from Baseline in EORTC QLQ- Non-Muscle-Invasive Bladder Cancer (NMIBC) 24 Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and 96
  EORTC QLQ-NMIBC24 is a 24-item questionnaire for evaluating the HRQoL of participants with NMIBC. The questionnaire is designed to supplement the QLQ-C30 and incorporates 6 multi-item scales (urinary symptoms, malaise, future worries, bloating and flatulence, sexual function and male sexual problems) and 5 single items (intravesical treatment issues, sexual intimacy, worries about risk of contaminating partner, sexual enjoyment, and female sexual problems). Ratings for each item range from 1 (not at all) to 4 (very much). Higher scores represent a high level of symptoms or problems, except for sexual function and sexual enjoyment, where a higher score represents a higher level of functioning.
Percentage of Participants With Meaningful Change From Baseline in EORTC-QLQ-C30 Scores | Weeks 12, 24, 36, 48, 60, 72, 84 and 96
  EORTC QLQ-C30 is a 30-item questionnaire for evaluating the health-related quality of life (HRQoL) of participants participating in cancer clinical studies. It includes 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea or vomiting), a global health status or HRQoL scale and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Ratings for each item range from 1 (not at all) to 4 (very much). Higher scores indicate greater functioning, better global health status, or more severe symptoms.
Percentage of Participants With Meaningful Change From Baseline in EORTC-QLQ-NMIBC24 Scores | Weeks 12, 24, 36, 48, 60, 72, 84 and 96
  EORTC QLQ-NMIBC24 is a 24-item questionnaire for evaluating the HRQoL of participants with NMIBC. The questionnaire is designed to supplement the QLQ-C30 and incorporates 6 multi-item scales (urinary symptoms, malaise, future worries, bloating and flatulence, sexual function and male sexual problems) and 5 single items (intravesical treatment issues, sexual intimacy, worries about risk of contaminating partner, sexual enjoyment, and female sexual problems). Ratings for each item range from 1 (not at all) to 4 (very much). Higher scores represent a high level of symptoms or problems, except for sexual function and sexual enjoyment, where a higher score represents a higher level of functioning.
Number of Participants with Overall Side Effects Measured by EORTC Question 168 (Q168) | Up to Week 96
  EORTC Q168 is a single item from the EORTC item library used to measure the overall impact of treatment side effects. Responses are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much." Higher score indicates greater impact.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (88):
- United States (18):
  - Colorado Clinical Research, Lakewood, Colorado
  - Georgia Urology, Atlanta, Georgia
  - Associated Urological Specialists, Chicago Ridge, Illinois
  - Urology of Indiana, Carmel, Indiana
  - Greater Boston Urology, Plymouth, Massachusetts
  - Comprehensive Urology, Royal Oak, Michigan
  - UroHealth Partners, Omaha, Nebraska
  - Dayton Physicians Network Urology, Centerville, Ohio
  - The Urology Group, Cincinnati, Ohio
  - Helios Clinical Research, LLC, Middleburg Heights, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - MidLantic Urology, Lancaster, Pennsylvania
  - University Of Pittsburgh Medical Center UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - The Conrad Pearson Clinic, Germantown, Tennessee
  - Urology Austin, Austin, Texas
  - Urology San Antonio PA dba USA Clinical Trials, San Antonio, Texas
- Argentina (5):
  - Hospital Sirio Libanes, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Investigaciones Clinico Moleculares (ICM), Caba
  - Centro Urologico Profesor Bengio, Córdoba
  - Sanatorio de la Mujer, Rosario
- Belgium (4):
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Maria Middelares, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Algemeen Ziekenhuis Delta, Roeselare
- Brazil (5):
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Hospital Regional do Cancer - Hospital de Esperança, Presidente Prudente
  - Fundacao Faculdade Regional De Medicina De Sao Jose Do Rio Preto, São José do Rio Preto
  - Fundacao Faculdade de Medicina Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
- China (7):
  - Peking University First Hospital, Beijing
  - The Third People's Hospital of Chengdu, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - Nanjing Drum Tower Hospital, Nanjing
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - The Second Hospital Of Tianjin Medical University, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
- France (6):
  - Institut Paoli Calmettes, Marseille
  - Hopital Saint Louis, Paris
  - CHU Pitie Salpetriere, Paris
  - Clinique de la Croix du Sud, Quint-Fonsegrives
  - CHP Saint Gregoire, Saint-Grégoire
  - Gustave Roussy, Villejuif
- Germany (6):
  - Universitaetsklinikum Koeln, Cologne
  - Marien hospital Herne, Herne
  - Klinikum Leverkusen gGmbH, Leverkusen
  - Universitaetsklinikum Mannheim, Mannheim
  - Studienpraxis Urologie Nurtingen, Nürtingen
  - Caritas-Krankenhaus St. Josef, Regensburg
- Greece (4):
  - General Hospital of Athens G Gennimatas, Athens
  - Laiko General Hospital of Athens, Athens
  - General Hospital Of Thessaloniki Papageorgiou, Thessaloniki
  - Athens Medical Center S A Interbalkan Medical Center of Thessaloniki, Thessaloniki
- Israel (6):
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - Cliniche Humanitas Gavazzeni, Bergamo
  - SPDC Villa Scassi, Genova
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Ospedale S. Maria Della Misericordia, Udine
- Japan (8):
  - Juntendo University Hospital, Bunkyō City
  - Funabashi Municipal Medical Center, Funabashi Shi
  - Hakodate Goryoukaku Hospital, Hakodate
  - St Marianna University Hospital, Kawasaki
  - Toho University Sakura Medical Center, Sakura
  - The Jikei University Hospital, Tokyo
  - Yokohama Municipal Citizen's Hospital, Yokohama
  - Yokohama City University Medical Center, Yokohama
- South Korea (5):
  - Chungbuk National University Hospital, Cheongju-si
  - Samsung Medical Center, Gangnam Gu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (5):
  - Hosp. Clinic de Barcelona, Barcelona
  - Hosp. Gral. Univ. de Castellon, Castellon
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp.Univ.Parc Tauli, Sabadell
- United Kingdom (5):
  - Hull University Teaching Hospitals NHS Trust, Cottingham
  - St Bartholomews Hospital, London
  - Southampton University Hospital, Southampton
  - Lister Hospital, Stevenage
  - Royal Marsden Hospital, Surrey

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency